CLINICAL TRIAL: NCT03538704
Title: Effect of Fertility-sparing Therapy of Early Endometrial Cancer
Acronym: ECFerSp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Peking University First Hospital (Other); Peking University Third Hospital (Other); Tianjin Medical University General Hospital (Other); Maternal and Child Health Hospital of Hubei Province (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018ECFerSp
Record Dates: First submitted 2018-03-14; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Endometrial Cancer; Fertility
Keywords: Endometrial cancer; Atypical hyperplasia; Fertility-preserving; Remission time; Recurrence; Pregnancy; Progesterone receptor
MeSH Terms: conditions — Endometrial Neoplasms; Recurrence | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BMI≥25 group with metformin (Experimental): Patients with BMI≥25kg/m2 in the experimental group are treated with medroxyprogesterone acetate (MPA) 0.25g/d plus metformin and are followed-up of baseline data, hormone levels,
  Interventions: Drug: Metformin
- BMI≥25 group without metformin (No Intervention): Patients with BMI≥25kg/m2 in the none intervention group are treated with MPA 0.25g/d alone and are followed-up of baseline data, hormone levels, and endometrial pathology every 3 months until 12 months.

INTERVENTIONS:
Drug: Metformin — Metformin is given to patients 1-1.5g/d.
  Arms: BMI≥25 group with metformin

SUMMARY:
The purpose of this study is to investigate the effect of Fertility-sparing Therapy of Early Endometrial Cancer.

DETAILED DESCRIPTION:
This is a prospective, multi center, open, randomized, controlled clinical trial. All endometrial cancer (EC) or atypical hyperplasia (AH) patients who met the fertility-sparing indications in the hospitals involved in this study were recruited. Then the investigators conducted assessment, treatment and follow up according to the standard procedure. General information, therapeutic regimen, side effects, oncological and pregnant results were collected for risk factors analysis.

ELIGIBILITY:
Inclusion Criteria:

* ages of no more than 40
* with a strong desire of fertility preservation
* International Federation of Gynecology and Obstetrics (FIGO) 2009 stage Ⅰa grade 1~2 with lesion confined in endometrium
* pathology expression of progestin receptors (PRs) and estrogen receptors

Exclusion Criteria:

* not eligible for pregnancy or delivery
* evidence of suspected extrauterine or distant metastasis
* complicated with any other malignancy
* severe medical complications
* contraindication of oral progestin
* uncontrolled epilepsy, central nervous system disease or mental disorder history in patients which Influence clinical research compliance judging by the researcher.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | through study completion, an average of 3 months
  Histologically shows absence of pathological hyperplasia or carcinoma.

SECONDARY OUTCOMES:
Pregnancy rate | through study completion, an average of 3 months
  Pregnancy test shows pregnancy after complete response.

OTHER OUTCOMES:
Recurrence rate | through study completion, an average of 3 months
  Pathology shows atypical hyperplasia or carcinoma again after complete response.

CONTACTS AND LOCATIONS:
Overall Officials: Jianliu Wang, Professor, Study Chair — Department of Obstetrics and Gynecology, Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gallos ID, Yap J, Rajkhowa M, Luesley DM, Coomarasamy A, Gupta JK. Regression, relapse, and live birth rates with fertility-sparing therapy for endometrial cancer and atypical complex endometrial hyperplasia: a systematic review and metaanalysis. Am J Obstet Gynecol. 2012 Oct;207(4):266.e1-12. doi: 10.1016/j.ajog.2012.08.011. Epub 2012 Aug 10. PMID 23021687